CLINICAL TRIAL: NCT02553031
Title: Application of MR-PET in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201403082MIND
Record Dates: First submitted 2015-09-10; First posted 2015-09-17 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
Keywords: Application of MR-PET
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: The imaging biomarkers determined by MR-PET — This study will explore the potential value in proper therapeutic decision and clinical outcome prediction by using integrated MR-PET system and advanced MR techniques in patients with colorectal cancer.

SUMMARY:
This study will explore the potential value in proper therapeutic decision and clinical outcome prediction by using integrated MR-PET system and advanced MR techniques in patients with colorectal cancer.

DETAILED DESCRIPTION:
This research expect that the image techniques and experience in this cancer group may be valuable and helpful for others. With advantage of MR-PET in better soft tissue delineation/functional information and less radiation dose than PET-CT, the ultimate goal in both research and clinical application is to establish new diagnostic standard and management guideline by MR-PET, which can further improve clinical outcome and disease prognosis in patients colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1: Patients with newly diagnosed colorectal cancers
2. Group 2: Patients with suspicious recurrent colorectal cancers

Exclusion Criteria:

1. Age <20 or >90 years old
2. Contraindication for MRI: claustrophobia or MR non-compatible devices
3. Contraindication for MR contrast medium: severe adverse reaction or impaired renal function (Cre > 2.0)
4. History of other malignancy
5. Prior arthroplasty of hip (may cause artifacts on MRI)
6. Pregnancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study. Patients with 50 newly diagnosed colorectal cancers and 50 patients with suspicious recurrent colorectal cancers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate at 1 year after surgery | 1 year

SECONDARY OUTCOMES:
The overall survival at 1 year after surgery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Fang Shih, M.D., Principal Investigator — Department of Medical Imaging, National Taiwan University Hospital.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan